CLINICAL TRIAL: NCT04144608
Title: A Phase II Study on Toripalimab Combined With Double Platinum Based Chemotherapy for as a Neoadjuvant Therapy for Initially Unresectable Non-driver Gene Mutation Non-small Cell Lung Cancer
Brief Title: Toripalimab Combined With Double Platinum-based Chemotherapy for Initially Unresectable NSCLC
Acronym: TOGATHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOGATHER
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Toripalimab NSCLC
MeSH Terms: interventions — toripalimab; Platinum Compounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Platinum-containing Dual-agent (Experimental): Toripalimab combined with platinum-containing dual-agent as a neoadjuvant Therapy for Non-small Cell Lung Cancer
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Nab-paclitaxel/pem +cisplatin +PD-1(Nab-paclitaxel260mg/m2 D1 Cisplatin 75mg/m2 D1 or carboplatin,determined by the investigator AUC)PD-1 200mg D1
  Other Names: platinum-based chemotherapy

SUMMARY:
The aim of the study was to investigate the efficacy of Toripalimab Combined with Double Platinum Based Chemotherapy for Initially Unresectable Non-driver Gene Mutation Non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
The aim of the study was to investigate the efficacy of Toripalimab Combined with Double Platinum Based Chemotherapy for Initially Unresectable Non-driver Gene Mutation Non-small Cell Lung Cancer. Other multiple Omics data will be analyzed to predict the MPR for treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have fully understood the trial and are willing to sign the informed consent form.
2. Ages between 18 years old to 70 years old, with no gender restrictions.
3. Previously untreated, histologically confirmed, potentially resectable stage IIIA-IIIB NSCLC (AJCC staging 8th edition); potentially resectable refers to patients with T3 or T4 primary lesions and positive N1 or N2 lymph nodes who are expected to be difficult to resect or require pneumonectomy after discussion by MDT (including surgery, imaging, anesthesia, and internal medicine).
4. Patients diagnosed with squamous cell carcinoma do not need genetic testing. If the test is positive for EGFR, ALK or ROS1, it is considered an exclusion criterion; if it is adenocarcinoma, genetic testing must include at least EGFR, ALK, and ROS1. The acceptable detection methods are ARMS or NGS, where NGS is a cFDA-approved test kit.
5. Measurable lesions according to Response Evaluation Criteria in Solid Tumors Version 1.1.
6. Before enrollment, 20 tissue sections (thickness 4-6 microns) must be submitted for biomarker evaluation (tumor tissue samples must be fresh or archived samples obtained within 3 months before enrollment; fresh tissue must be core needle biopsy, excision, or incision biopsy specimens).
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
8. Good organ function:
9. Hematology: absolute neutrophil count (ANC) ≥ 1500/μL; platelets ≥ 100,000/μL; hemoglobin ≥ 9.0g/dL or ≥ 5.6 mmol/L;
10. Kidney: serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cock-Gault formula);
11. Liver: Total bilirubin ≤ 1.5 × ULN or direct bilirubin within normal limits for subjects with total bilirubin levels > 1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN;
12. Endocrine system: Thyroid stimulating hormone (TSH) within normal limits. Note: If TSH is not within the normal range at baseline, the subject may still meet the inclusion criteria if T3 and free T4 are within the normal range;
13. Coagulation function: International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, except for subjects who are receiving anticoagulant therapy, as long as PT or aPTT is within the intended use range of the anticoagulant drug; (1)Cardiac function test: Baseline electrocardiogram shows no PR interval prolongation or atrioventricular block;
14. Total lung function is adequate to sustain the planned lung resection, as assessed by the surgeon.

Women must agree to use contraceptive measures (such as intrauterine devices (IUDs), birth control pills or condoms) during the study and within 6 months after the study ends; serum or urine pregnancy tests must be negative within 7 days before study enrollment, and must not be breastfeeding patients; men must agree to use contraceptive measures during the study and within 6 months after the study ends.

Exclusion Criteria:

1. Histopathological identification is neuroendocrine carcinoma or sarcomatoid tumor.
2. Resectable disease in the early stage.
3. Subjects with known EGFR mutations or ALK, ROS1 translocations, and subjects with non-squamous cell carcinoma need to clarify the EGFR, ALK and ROS1 mutation status.
4. Early-stage NSCLC who have received prior systemic anticancer therapy, including investigational drugs.
5. History of (non-infectious) pneumonitis/interstitial lung disease requiring steroids, or current pneumonitis/interstitial lung disease requiring steroids.
6. Known history of active tuberculosis.
7. Known active infection requiring systemic therapy.
8. Subjects with any known or suspected autoimmune disease or immunodeficiency, except patients with a history of hypothyroidism who do not require hormone therapy or are receiving physiological doses of hormone replacement therapy; subjects with stable type 1 diabetes with controlled blood glucose.
9. Subjects with active hepatitis B (defined as a positive result of hepatitis B virus surface antigen [HBsAg] test during the screening period and a HBV-DNA test value higher than the upper limit of the normal value of the laboratory department of the research center) or hepatitis C (defined as a positive result of hepatitis C virus surface antibody [HCsAb] test during the screening period and a positive HCV-RNA test result).
10. Known human immunodeficiency virus (HIV) infection (known HIV antibody positive).
11. Live vaccines within 30 days prior to first dose. Including but not limited to the following: mumps, rubella, measles, varicella/zoster (chickenpox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccines (inactivated virus vaccines are permitted).
12. Have grade ≥ 2 peripheral neuropathy.
13. Patients who have received previous treatment with PD-1/PD-L1 drugs or another drug targeting T cell receptors (e.g. CTLA-4, OX-40, etc.).
14. Patients with any severe and/or uncontrolled illness:

(1)patients with unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; patients with poorly controlled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);.

(2)active or uncontrolled severe infection; (3)liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis; (4)poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L); (5)patients with urine routine test indicating urine protein ≥ ++ and confirmed 24-hour urine protein quantitative > 1.0g; (6)patients with a history of psychotropic drug abuse and unable to quit or with mental disorders; (7)Use of immunosuppressive drugs within 2 weeks before the first study drug treatment, excluding topical glucocorticoids or systemic glucocorticoids not exceeding 10 mg/day of prednisone or other glucocorticoids at equivalent doses.

15.Pregnant or lactating women. 16.Prisoners who are illegally imprisoned or detained for reasons other than mental illness or physical illness (such as infectious diseases).

17.Patients with bleeding tendencies (eg., active peptic ulcers) or who are treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogs.

18.History of study drug allergy. 19.According to the researcher's judgment, patients with concomitant diseases that seriously endanger patient safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
R0 surgical resection rate | Approximately 1 years
  No residual ratio under the microscope after surgical resection

SECONDARY OUTCOMES:
ORR | Approximately 2 years
  To measure the patients's overall response rate
Major Pathological Response (MPR) rate | Approximately 2 years
  defined as noadjuvant therapy-induced tumor regression in pathologically residual tumor cells <10%
Complete Response (pCR) rate | Approximately 2 years
  Defined as non-adjuvant therapy-induced tumor regression in absence of pathologically residual tumor cells
Event-Free Survival (EFS) | Approximately 2 years
  Defined as the time from the first dose treatment to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death.
Disease-Free Survival (DFS) | Approximately 2 years
  Defined as the time from surgery to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death.
Overall Survival (OS) | Approximately 2 years
  Defined as the time from the first dose treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Z MD, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zeng L, Yan H, Jiang W, Qin H, Dai J, Zhang Y, Wei S, Chen S, Liu L, Xiong Y, Yang H, Li Y, Wang Z, Deng L, Xu Q, Peng L, Zhang R, Fang C, Chen X, Deng J, Wang J, Li T, Liu H, Zhang G, Yang N, Zhang Y. Toripalimab plus platinum-doublet chemotherapy as perioperative therapy for initially unresectable NSCLC: An open-label, phase 2 trial. Med. 2025 Jun 13;6(6):100574. doi: 10.1016/j.medj.2025.100574. Epub 2025 Jan 31. PMID 39892382